CLINICAL TRIAL: NCT05822687
Title: Promoting Effective Coping by Children Exposed to Post-divorce Interparental Conflict to Reduce Risk for Mental Health Problems
Brief Title: Factorial Optimization Trial to Test Effects of Coping Intervention Components
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Karey O'Hara, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00016078; K01MH120321 (NIH)
Record Dates: First submitted 2023-02-17; First posted 2023-04-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Depression; Coping Skills; Emotional Problem
Keywords: optimization; parental divorce/separation; interparental conflict; adaptive coping; child mental health
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Education (Experimental): Participants will complete an educational digital module and no skills-based digital modules.
  Interventions: Behavioral: Education
- Education + Reappraisal (Experimental): Participants will complete an educational digital module and a skills-based digital module that teaches reappraisal coping.
  Interventions: Behavioral: Education; Behavioral: Reappraisal Coping
- Education + Distraction (Experimental): Participants will complete an educational digital module and a skills-based digital module that teaches distraction coping.
  Interventions: Behavioral: Education; Behavioral: Distraction Coping
- Education + Relaxation (Experimental): Participants will complete an educational digital module and a skills-based digital module that teaches relaxation coping.
  Interventions: Behavioral: Education; Behavioral: Relaxation Coping
- Education + Reappraisal + Distraction (Experimental): Participants will complete an educational digital module and two skills-based digital modules, one that teaches reappraisal coping and one that teaches distraction coping.
  Interventions: Behavioral: Education; Behavioral: Reappraisal Coping; Behavioral: Distraction Coping
- Education + Reappraisal + Relaxation (Experimental): Participants will complete an educational digital module and two skills-based digital modules, one that teaches reappraisal coping and one that teaches relaxation coping.
  Interventions: Behavioral: Education; Behavioral: Reappraisal Coping; Behavioral: Relaxation Coping
- Education + Distraction + Relaxation (Experimental): Participants will complete an educational digital module and two skills-based digital modules, one that teaches distraction coping and one that teaches relaxation coping.
  Interventions: Behavioral: Education; Behavioral: Distraction Coping; Behavioral: Relaxation Coping
- Education + Reappraisal + Distraction + Relaxation (Experimental): Participants will complete an educational digital module and three skills-based digital modules, one that teaches reappraisal coping, one that teaches distraction coping, and one that teaches relaxation coping.
  Interventions: Behavioral: Education; Behavioral: Reappraisal Coping; Behavioral: Distraction Coping; Behavioral: Relaxation Coping

INTERVENTIONS:
Behavioral: Education — This is a constant component; all participants will get a psychoeducation digital module.
Behavioral: Reappraisal Coping — This digital module will teach reappraisal coping skills.
  Arms: Education + Reappraisal; Education + Reappraisal + Distraction; Education + Reappraisal + Distraction + Relaxation; Education + Reappraisal + Relaxation
Behavioral: Distraction Coping — This digital module will teach distraction coping skills.
  Arms: Education + Distraction; Education + Distraction + Relaxation; Education + Reappraisal + Distraction; Education + Reappraisal + Distraction + Relaxation
Behavioral: Relaxation Coping — This digital module will teach relaxation coping skills.
  Arms: Education + Distraction + Relaxation; Education + Reappraisal + Distraction + Relaxation; Education + Reappraisal + Relaxation; Education + Relaxation

SUMMARY:
This study will identify components for inclusion in a coping intervention package to reduce mental health problems among children exposed to high interparental conflict after parental separation/divorce. Reappraisal, distraction, and relaxation coping strategies are related to fewer mental health problems among children, making intervention components based on these strategies key candidates for inclusion in an optimized coping intervention. The primary aim is to experimentally assess the main and interactive effects of three digital intervention coping components (reappraisal, distraction, relaxation) on children's coping efficacy, emotional security, and internalizing and externalizing problems. Secondary aims are to assess indirect effects of the intervention components on children's coping efficacy, emotional security, and internalizing and externalizing problems through their cognitive, emotional, and behavioral reactions to post-separation/divorce interparental conflict events.

DETAILED DESCRIPTION:
A randomized and counterbalanced 2x2x2 factorial trial (N = 144 children, ages 9-12) will be conducted to assess the individual effects of the three digital coping intervention components. The three components to be tested will be: (1) Reappraisal (No vs. Yes), (2) Distraction (No vs. Yes), (3) Relaxation (No vs. Yes). Components that meet a priori thresholds for meaningful change will be combined to form an intervention package that will be evaluated in a subsequent randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* child between ages 9-12 whose parents are separated or divorced
* child and one parent are fluent in English
* a parent with sufficient contact (i.e., at least 4 overnights and/or 12 daytime visits per month) with child who is willing to complete study assessments and has legal right to give permission for the child to participate in research
* child-report of high exposure to IPC (mean Z score ≥ 40th percentile on the two child report measures of IPC; score standardization based on data from 559 youth whose parents participated in an experimental parenting program)
* elevated internalizing or externalizing problems (T score in the borderline clinical range according to either child or parent report on the BPM).

Exclusion Criteria:

* in active therapy
* score ≥ 99th percentile on either internalizing and externalizing problems subscale
* endorse suicidality (will be ineligible for the study and referred for treatment)

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2023-02-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
interparental emotional security | pretest at study entry
  Security in the Interparental Subsystem Scale - Short Form (SIS-SF; Holt et al., 2020) 17 items rated on 4 point scale (0 = not at all true, 3 = very true for me) higher scores indicate better outcome
interparental emotional security | posttest at one month after completion of the last assigned intervention module
  Security in the Interparental Subsystem Scale - Short Form (SIS-SF; Holt et al., 2020) 17 items rated on 4 point scale (0 = not at all true, 3 = very true for me) higher scores indicate better outcome
interparental emotional security | follow-up at 3 months after completion of the last assigned intervention module
  Security in the Interparental Subsystem Scale - Short Form (SIS-SF; Holt et al., 2020) 17 items rated on 4 point scale (0 = not at all true, 3 = very true for me) higher scores indicate better outcome
family emotional security | pretest at study entry
  Security in the Family System Scale (SIFS; Forman & Davies, 2005) 24 items rated on 4 point scale (0 = completely disagree, 3 = completely agree).
  higher scores indicate better outcome
family emotional security | posttest at one month after completion of the last assigned intervention module
  Security in the Family System Scale (SIFS; Forman & Davies, 2005) 24 items rated on 4 point scale (0 = completely disagree, 3 = completely agree).
  higher scores indicate better outcome
family emotional security | follow-up at 3 months after completion of the last assigned intervention module
  Security in the Family System Scale (SIFS; Forman & Davies, 2005) 24 items rated on 4 point scale (0 = completely disagree, 3 = completely agree).
  higher scores indicate better outcome
coping efficacy | pretest at study entry
  Coping Efficacy Scale (CES; Sandler et al., 2000) 7 items rated on 4 point scale (0 = not at all, 3 = very) higher scores indicate better outcome
coping efficacy | posttest at one month after completion of the last assigned intervention module
  Coping Efficacy Scale (CES; Sandler et al., 2000) 7 items rated on 4 point scale (0 = not at all, 3 = very) higher scores indicate better outcome
coping efficacy | follow-up at 3 months after completion of the last assigned intervention module
  Coping Efficacy Scale (CES; Sandler et al., 2000) 7 items rated on 4 point scale (0 = not at all, 3 = very) higher scores indicate better outcome
internalizing problems | pretest at study entry
  Brief Problem Monitor (BPM; parent and child report) 6 items rated on a 3 point scale (0= not true, 2 = very true) higher scores indicate worse outcome
internalizing problems | posttest at one month after completion of the last assigned intervention module
  Brief Problem Monitor (BPM; parent and child report) 6 items rated on a 3 point scale (0= not true, 2 = very true) higher scores indicate worse outcome
internalizing problems | follow-up at 3 months after completion of the last assigned intervention module
  Brief Problem Monitor (BPM; parent and child report) 6 items rated on a 3 point scale (0= not true, 2 = very true) higher scores indicate worse outcome
externalizing problems | pretest at study entry
  Brief Problem Monitor (BPM; parent and child report) 7 items rated on a 3 point scale (0= not true, 2 = very true) higher scores indicate worse outcome
externalizing problems | posttest at one month after completion of the last assigned intervention module
  Brief Problem Monitor (BPM; parent and child report) 7 items rated on a 3 point scale (0= not true, 2 = very true) higher scores indicate worse outcome
externalizing problems | follow-up at 3 months after completion of the last assigned intervention module
  Brief Problem Monitor (BPM; parent and child report) 7 items rated on a 3 point scale (0= not true, 2 = very true) higher scores indicate worse outcome

SECONDARY OUTCOMES:
Cognitive appraisals - conflict specific | daily (6 weeks)
  SIS-SF Internal Representations subscale (Holt et al., 2020; 6 items)
Cognitive appraisals - general | daily (6 weeks)
  Threat and Worry Appraisal Scale (TWAS; Sheets et al., 1996; 6 items)
Emotional distress | daily (6 weeks)
  SIS-SF Emotional Reactivity subscale (Holt et al., 2020; 3 items)
Physiological arousal | daily (6 weeks)
  Responses to Stress Questionnaire for Parent Conflict Involuntary Engagement subscale (RSQ-PC; Connor-Smith et al., 2000; 3 items)
Coping behaviors - conflict specific | daily (6 weeks)
  SIS-SF Involvement subscale (Holt et al., 2020; 3 items)
Coping behaviors - general | daily (6 weeks)
  RSQ-PC primary control, secondary control, and disengagement coping subscales (Connor-Smith et al., 2000; 15-18 items).

CONTACTS AND LOCATIONS:
Overall Officials: Karey L O'Hara, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Study results will be shared through presentations at conferences and submissions in peer-reviewed journals. In addition, after taking all steps necessary to minimize possible re-identification of confidential data, I will make data, codebooks, and analysis scripts available to appropriate parties to verify findings and conclusions.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: one year post data collection
Access Criteria: qualified researchers who have gained IRB approval and pre-registered their analyses